CLINICAL TRIAL: NCT04302935
Title: Pain & Expert: Global Pain-assessment: a Prospective Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Prof. dr., Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: P&E
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic pain patients
  Interventions: Other: Global pain-assessment

INTERVENTIONS:
Other: Global pain-assessment — Global pain-assessment, based on the ICF framework

SUMMARY:
Full assessment of chronic pain patients based on the ICF-model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain for at least 3 months
* Age => 18 years
* Patient has been informed of the study procedures and has given written informed consent

Exclusion Criteria:

* Healthy patients or patients with acute pain.
* Addiction to drugs, alcohol (>5 units per day)
* Evidence of an active disruptive psychiatric disorder that may impact perception of pain, and/or ability to evaluate treatment outcome as determined by investigator
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a global pain-assessment (i.e. practical use) | at the time of the assessment: one day (cross-sectional)

SECONDARY OUTCOMES:
norm values for chronic pain patients on all aspects of the global pain-assessment will be reported (i.e. descriptives) | at the time of the assessment: one day (cross-sectional)
  Reporting of norm values on the different aspects of the ICF framework in patients with chronic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium